CLINICAL TRIAL: NCT06929351
Title: Effect of Otago Exercise Program in Comparison With Dual Task Training on Balance and Postural Control in Elderly Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/48
Record Dates: First submitted 2024-12-06; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Postural Balance; Posture; Aged; Exercise Therapy; Fall Prevention; Muscle Strength; Cognition
Keywords: Otago exercise program; dual task training; balance; postural control; functional mobility; risk of fall; older adults; berg balance scale; TUG; dynamic gait index; FES-I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago exercise group (Experimental): Otago exercise program consist of strengthening exercise of lower limb muscles and along with balance exercises. Knee flexors, knee extensors and hip abductors, which are particularly important or functional movements and walking. Ankle dorsiflexor and plantar flexor muscles, which are particularly important for recovering balance. Ankle cuff weights provide resistance to the knee flexors, knee extensors and hip abductors; the ankle dorsiflexors and plantar flexors are strengthened using body weight alone. The balance exercises are dynamic as well as static. They can help to maintain balance, postural control and functional mobility.
  The program was designed specifically to prevent falls. It consists of a set of leg muscle strengthening and balance retraining exercises progressing in difficulty, and a walking plan. The exercises are individually prescribed and increase in difficulty during a series of visits under a trained instructor. ankle cuff weights (starting at 1kg) t
  Interventions: Procedure: otago exercise
- Dual task group (Experimental): Dual task training (DTT) is an intervention that involves performing two tasks simultaneously, typically a motor task (e.g., walking, standing) and a cognitive task (e.g., solving a mental puzzle, counting). The aim is to improve balance, postural control, functional mobility, and cognitive function, which are crucial for reducing the risk of falls among older adults. As people age, they experience declines in several areas, including: Reduced muscle strength, flexibility, and coordination make movements like walking or maintaining balance more difficult, Declines in attention, memory, and executive functions (e.g., problem-solving, decision- making) can make it challenging to focus on multiple things at once. For older adults, this dual tasking can increase the risk of imbalance and falls. DTT aims to improve older adults' ability to manage these simultaneous demands, making daily life safer and more manageable. Dual task training focuses on performing a motor task and a c
  Interventions: Procedure: Dual task exercise

INTERVENTIONS:
Procedure: otago exercise — Otago exercise program group 40 min/ thrice a week/ 8 weeks
  1st week strengthening of knee flexors( prone lying), extensors ( in sitting) ,abductors( in standing) with 1-2 kg ankle cuff. Dorsi flexors, planter flexors(in standing on weight)/ hold 5-10 sec 5 reps/ 2 sets 2nd week Strengthening same as week 1 balance exercises.Knee bending( standing),tandem stance,sit to stand / with support/ 5-10 reps/2 sets 3rd week strengthening of all above Ms group with increase weight 2-3 kg ankle cuff or participant (The exercises are of moderate intensity; the person should not get unduly tired) balance exercise as 2nd week 4th week strengthening exs as in 3rd week balance exs: Knee bending, tandem stance( without support), forward walk,walking and turning around, side walk, one leg stand,sit to stand, stair climb( all with support)/5-10 reps 5th week strengthening exs of above ms group increase either weight 3-4 kg or repetitions 10-15 or hold time 10-15 sec 6th week strengthening same as 5
  Arms: Otago exercise group
Procedure: Dual task exercise — Balance exercises and secondary cognitive task simultaneously 40 min/ thrice a week/ 8 weeks
  1. st week Balance exercises: Narrow-base standing on the floor (firm surface) with eyes open and closed, Tandem standing on the floor with eyes open and closed, Single-leg standing on the floor with eyes open and closed, Wide-base walking on the floor, Chair sitting to standing transfer Cognitive tasks: Naming a group of cities; foodstuff; boy names; or girl names starting with A,I, S, and T sounds/ 3 trails
  2. nd week Balance exercise: Narrow-base standing on the floor with open eyes while moving arms, Forward lunge standing on the floor with eyes open, Narrow-base walking on the floor, keeping balance while sitting on a ball and moving arms in different directions Cognitive task: Backward counting from 50,Count by multiple(3,6,9…….)/3trails Week 3 Balance exercises: Narrow-base standing on a foam with eyes open and closed, Tandem standing on a foam with eyes open and closed, Backward walking on
  Arms: Dual task group

SUMMARY:
Balance and postural control are major concerns in reduction of risk of fall among older adults. Otago Exercise Program and dual task training program are commonly used approaches to improve balance, functional mobility and postural control. However, limited studies have compared the efficacy of Otago Exercise Program and dual task training program in improving balance and functional mobility. One-third to one-half of the population over age 60 reports injuries due to fall because of the high incidence of balance and mobility disorders in older adults, interventions are necessary that optimize the performance of balance- and mobility-related activities among older adults. The aim of the current study to find out better intervention which will benefit the clinicians and physiotherapists in clinical decision making of managing the geriatric population, suffering fear of fall, going to effect on their daily livings, with evidence.

DETAILED DESCRIPTION:
Objective of study:

* To determine the effect of Otago Exercise Program in comparison with Dual task training on balance in elderly population.
* To determine the effect of Otago Exercise Program in comparison with Dual task training on functional mobility in elderly population.
* To determine the effect of Otago Exercise Program in comparison with Dual task training on postural control in elderly population.
* To determine the effect of Otago Exercise Program in comparison with Dual task training on reduction the fear of fall in elderly population. Significance of study
* The study will be going to highlight whether healthy older adults who perform Otago exercise program would show significant improvement on balance and postural control in comparison with dual task training program.
* Through this research medical professionals may identify the best treatment protocol in reduction of fear of fall among older adults.
* This study will helpful for the physiotherapists in clinical decision making of managing the geriatric population, suffering fear of fall, going to effect on their daily livings, with evidence.
* It will provide research data for further study and fill the research gap. Alternate hypothsis
* There will be statistically significant difference between Otago Exercise Program in comparison with Dual task training on balance in elderly population. (p<0.05)
* There will be statistically significant difference between Otago Exercise Program in comparison with Dual task training on postural control in elderly population. (p<0.05).
* There will be statistically significant difference between Otago Exercise Program in comparison with Dual task training on fear of fall in elderly population. (p<0.05)
* There will be statistically significant difference between Otago Exercise Program in comparison with Dual task training on functional mobility in elderly population (p<0.05).

Null hupothesis

* There will be no statistically significant difference between Otago Exercise Program in comparison with Dual task training on balance in elderly population. (p>0.05)
* There will be no statistically significant difference between Otago Exercise Program in comparison with Dual task training on postural control in elderly population. (p>0.05)
* There will be no statistically significant difference between Otago Exercise Program in comparison with Dual task training on fear of fall in elderly population. (p>0.05)
* There will be no statistically significant difference between Otago Exercise Program in comparison with Dual task training on functional mobility in elderly population. (p>0.05)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* both male and female,
* Older adults who are functionally independent,
* Can walk independently or with assistive devices will be considered typical healthy,
* Can sit to stand with or without support,
* Mini-mental status examination ≥ 24.

Exclusion Criteria:

* history of fracture especially in the lower limb,
* major cognitive issues (e.g. Alzheimer's disease, dementia),
* major orthopedic problems (e.g. lower limb fractures, amputation),
* neurological disease (e.g. stroke, Parkinson disease) or any other comorbidities that restrict mobility
* marked impairment of visual and vestibular function.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Balance | 8 weeks
  Berg balance scale is used to assess static and dynamic balance having 14 balance tasks Scoring: 5-point ordinal scale (graded 0-4) , Max score = 56 41-56 = low fall risk, 21-40 = medium fall risk, 0 -20 = high fall risk Perform at the start of treatment protocol, after 4 weeks and at the end of intervention
Postural Control | 8 weeks
  tool used for assessment of postural control is Dynamic gait index. It includes eight items, A four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function.
  Total Score = 24. < 19/24 = predictive of falls in the elderly, > 22/24 = safe ambulators
risk of fall | 8 weeks
  tool used to assess fall risk is FES-I. 16 items Questionnaire. individuals are instructed to score their concern of falling during an activity on a 4 point Likert scale with 1 as not concerned at all and 4 as very concerned. The item scores are summed up to obtain a total of 64. ≤ 16= no concern about falling > 16= concern about falling
Functional Mobility | 8 weeks
  tool used for assessment of functional mobility is Timed Up And Go. Uses 1 practice/3 trials for average score. If the participant perform it with in 10 sec will be consider normal, > 10 second= impaired functional mobility lead to moderate to high risk of fall.
Functional Mobility Strength | 8 weeks
  Tool used for assessment of functional mobility strength is Sit to stand 30 sec: The score is the total number of stands with in 30 sec. For men and women above 60 years normal average score is 15 and 12 respectively below average score indicates a risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan